CLINICAL TRIAL: NCT04485715
Title: Application of Artificial Intelligence in Colorectal Polypectomy
Brief Title: Application of AI in Polypectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, gastroenterology professor of Qilu Hospital, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020SDU-QILU-0714
Record Dates: First submitted 2020-07-14; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps | interventions — Intelligent Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-aided group (Experimental)
  Interventions: Other: AI system
- control group (No Intervention)

INTERVENTIONS:
Other: AI system — The real-time assistance of AI system
  Arms: AI-aided group

SUMMARY:
The aim of this study was to assess the performance of AI system in polypectomy

ELIGIBILITY:
Inclusion Criteria:

* to undergo colorectal polypectomy;
* agree to give written informed consent

Exclusion Criteria:

* patients with the contraindications to colorectal polypectomy;
* patients with a history of inflammatory bowel disease (IBD), CRC, colorectal surgery;
* patients with high suspicion of polyposis syndromes, IBD and typical advanced CRC;
* patients refused to participate in the trial;
* the procedure cannot be completed due to stenosis, obstruction, huge occupying lesions, or solid stool;
* the procedure have to be terminated due to complications of anaesthesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-21 (Estimated); Primary Completion 2021-07-21 (Estimated); Study Completion 2021-09-21 (Estimated)

PRIMARY OUTCOMES:
polypectomy time | 12 months
  the time for detection in polypectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China